CLINICAL TRIAL: NCT05808556
Title: Efficacy and Safety of Sticker Pad Containing Essential Oil in Volunteer With High Blood Pressure
Brief Title: Sticker Pad Containing Essential Oil in Volunteer With High Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Pornanong Aramwit, Pharm.D., Ph.D, Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC 21233-20
Record Dates: First submitted 2023-03-14; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: High Blood Pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sticker pads containing lavender and ylang ylang oil (Experimental): The subjects in the sticker pad group attached an sticker pad (0.3% lavender oil and 0.7% ylang ylang oil) to their shirt, close to the right side of the neck, for 14 days
  Interventions: Device: Sticker pads containing lavender and ylang ylang oil
- Placebo group (Placebo Comparator): The placebo group attached a sticker pad without lavender and ylang ylang oil to their shirt, close to the right side of the neck, for 14 days.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Sticker pads containing lavender and ylang ylang oil — The sticker pad group attached an sticker pad (0.3% lavender oil and 0.7% ylang ylang oil) to their shirt, close to the right side of the neck, for 14 days,
  Arms: Sticker pads containing lavender and ylang ylang oil
Device: Placebo — The placebo group attached a sticker pad without lavender and ylang ylang oil to their shirt, close to the right side of the neck, for 14 days.
  Arms: Placebo group

SUMMARY:
The aims of the study were to evaluate efficacy and safety of the sticker pads containing lavender and ylang ylang oil in high blood pressure volunteers

DETAILED DESCRIPTION:
High blood pressure volunteers were divided into the sticker group or the placebo group. The volunteers attached the pad to their shirt for 3, 7, 10, and 14 days. Blood pressure, pulse rate, adverse reactions, and satisfaction were investigated.

ELIGIBILITY:
Inclusion Criteria:

* age more than 18 years
* systolic blood pressure of more than 130 mmHg but less than 160 mmHg or diastolic blood pressure more than 80 mmHg but less than 100 mmHg
* no hypertensive medicine
* no dermatological diseases, immunocompromised diseases, seizures, asthma, or respiratory diseases

Exclusion Criteria:

* an unstable condition of other diseases
* olfactory problems
* pregnancy
* lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | 14 days
  Measure systolic blood pressure in mmHg
Diastolic blood pressure | 14 days
  Measure diastolic blood pressure in mmHg
Pulse rate | 14 days
  Measure pulse rate in beats/minutes

SECONDARY OUTCOMES:
adverse reactions of the respiratory tract, skin, gastrointestinal tract, eye, and central nervous system | 14 days
  Using a score of 0 to 3, following an increase of severity
Satisfaction of the product | 14 days
  Using a visual analogue scale, 0 means not satisfied, 10 means very satisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Chulalongkorn Hospital, Bangkok, Thailand